CLINICAL TRIAL: NCT06363695
Title: Implementing the Adapted Parenting Program, SafeCare Kenya, to Reduce Noncommunicable Disease Burden: Building Community Health Volunteers' Capacity to Support Parents With Young Children
Brief Title: Building Community Health Volunteers' Capacity to Support Parents With Young Children With SafeCare Kenya
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Georgia State University (Other); Africa Institute of Mental and Brain Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 131-22; 1R01HD112043-01 (NIH)
Record Dates: First submitted 2024-03-20; First posted 2024-04-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-04

CONDITIONS: Child Maltreatment; Parenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care as Usual (Active Comparator): Community Health Volunteers will continue their usual services with families. This is typically done on a monthly basis focused on physical health needs of the mother and/or child.
  Interventions: Other: Care as Usual by Community Health Volunteers
- SafeCare Kenya In-Person (Experimental): Community Health Volunteers randomized to SafeCare Kenya will be trained to deliver this program either virtually or in-person. The Community Health Volunteer's families enrolled in the study will be randomized to receive the program either virtually or in-person. For in-person families, the Community Health Volunteer will deliver the session in the mother's home. The SafeCare Kenya curriculum will be the same in both the virtual and in-person.
  Interventions: Behavioral: SafeCare Kenya
- SafeCare Kenya Virtual (Experimental): Community Health Volunteers randomized to SafeCare Kenya will be trained to deliver this program either virtually or in-person. The Community Health Volunteer's families enrolled in the study will be randomized to receive the program either virtually or in-person. For in-person families, the Community Health Volunteer will deliver the session via a virtual platform (e.g., Zoom). The SafeCare Kenya curriculum will be the same in both the virtual and in-person.
  Interventions: Behavioral: SafeCare Kenya

INTERVENTIONS:
Behavioral: SafeCare Kenya — Adapted from SafeCare, this is a strengths-based program for parents with children ages 18 months through age 5, teaching parents skills and knowledge in three areas: 1) parent-child interactions, 2) child health, and 3) home safety.
  Other Names: SafeCare
  Arms: SafeCare Kenya In-Person; SafeCare Kenya Virtual
Other: Care as Usual by Community Health Volunteers — Community Health Volunteers support families with children up to age 5 around the physical health needs of family members, including delivering key health messages (e.g., importance of immunizations); treating minor injuries and illnesses; identifying/treating/referring common childhood illnesses (e.g., diarrhea, malaria); conducting home visits to evaluate the home environment and discuss improvements; and encouraging care at home and appropriate health seeking behaviors. These support services are not highly structured but rather tailored to the needs of each family.
  Arms: Care as Usual

SUMMARY:
The goal of this clinical trial is to implement and examine the impact of SafeCare Kenya, an adapted parenting program, to improve parents' skills and knowledge related to the care of their children between the ages of 18 months and 5 years old. The main questions it aims to answer are:

* Will SafeCare Kenya improve child and parent outcomes?
* Is virtual delivery as effective as in-person delivery of SafeCare Kenya?
* Is SafeCare Kenya feasible to deliver by community health volunteers?

Mothers will:

* Complete study assessments at three timepoints: baseline, 6 months and 18 months
* Mothers in the SafeCare Kenya group will receive the program from their community health volunteer

Researchers will compare SafeCare Kenya to care as usual by community health volunteers to see if SafeCare Kenya families show improvements in parent interaction skills, safety and health knowledge, potential for child abuse, child behavior problems, child injuries, parenting stress, and child and parent quality of life.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all community health volunteers consented to the study will be randomized to continue their usual services with families or be trained to deliver SafeCare Kenya to add to their usual services with families. All community health volunteers will inform their eligible families about the study and share with the research team mothers who express interest in the study. After being informed about the study and potential risks, all mothers giving informed consent will complete a baseline assessment, along with a 6 month and 18 month follow up assessment. Mothers whose community health volunteer is assigned to the SafeCare Kenya program will receive the program from their community health volunteers. All SafeCare Kenya mothers will be randomized to receive the program either in-person or virtually. Trainers and Stakeholders will provide information about their involvement in the project.

ELIGIBILITY:
Parents Inclusion Criteria:

* being the female primary caregiver
* at least 18 years old of age
* at least one child between 18 months and age 5
* reside in Kibera
* have ability to participate virtually (i.e., owns a smart phone) in English or Swahili.

Parent Exclusion Criteria:

* younger than 18 years old
* unable to participate in English or Swahili
* does not own smart phone to participate in virtual sessions.

CHV Inclusion Criteria:

* 18 years or older
* able to participate in English or Swahili
* has ability to participate virtually (i.e., owns a smart phone)
* female community health volunteer who is affiliated with one of the project's agencies in Kibera

CHV Exclusion Criteria:

* younger than 18 years old
* not able to participate in English or Swahili
* does not have a smart phone
* is not female
* is not a community health volunteer affiliated with one of the project's agencies

Trainer Inclusion Criteria:

* 18 years or older
* able to participate in English and Swahili
* trained as a SafeCare trainer

Trainer Exclusion Criteria:

* younger than 18 years old
* not able to participate in English and Swahili
* not trained as a SafeCare Trainer

Stakeholder Inclusion Criteria:

* 18 years or older
* able to participate in English
* involved in the project as a stakeholder

Stakeholder Exclusion Criteria:

* younger than 18 years old
* not able to participate in English
* not a stakeholder for this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in score on Child Planned Activities Training (cPAT) at 6 months | Baseline and 6 months
  The SafeCare Kenya form, cPAT, will be used to assess positive parent interaction skills. It is an observation of the 10 targeted skills in the SCK program. The assessor will virtually observe 1 play interaction. They rate parents using a minus when no skills present, check when some, and check plus when all aspects of the skill are present.
Change from Baseline in score on Child Planned Activities Training (cPAT) at 18 months | Baseline and 18 months
  The SafeCare Kenya form, cPAT, will be used to assess positive parent interaction skills. It is an observation of the 10 targeted skills in the SCK program. The assessor will virtually observe 1 play interaction. They rate parents using a minus when no skills present, check when some, and check plus when all aspects of the skill are present.
Change from Baseline in scores on Parenting Young Children (PARYC) at 6 months | Baseline and 6 months
  21 items assess a range of positive parenting practices, such as praise/rewards, planning for transitions, and providing choices among other practices. Items are summed to create an overall parent-child interaction score.
Change from Baseline in scores on Parenting Young Children (PARYC) at 18 months | Baseline and 18 months
  21 items assess a range of positive parenting practices, such as praise/rewards, planning for transitions, and providing choices among other practices. Items are summed to create an overall parent-child interaction score.
Change from Baseline in score on How to Keep your Child Safe and Healthy Quiz at 6 months | Baseline and 6 months
  The Quiz will be used to assess knowledge and skills related to the health and safety portions of the SafeCare Kenya intervention.
Change from Baseline in score on How to Keep your Child Safe and Healthy Quiz at 18 months | Baseline and 18 months
  The Quiz will be used to assess knowledge and skills related to the health and safety portions of the SafeCare Kenya intervention.
Change from Baseline in score on Brief Child Abuse Potential Inventory (BCAPI) at 6 months | Baseline and 6 months
  The BCAPI assesses parents' potential to engage in child maltreatment related behaviors. The 24 risk scale items are summed to create a total abuse potential score, with higher scores indicating higher abuse potential.
Change from Baseline in score on Brief Child Abuse Potential Inventory (BCAPI) at 18 months | Baseline and 18 months
  The BCAPI assesses parents' potential to engage in child maltreatment related behaviors. The 24 risk scale items are summed to create a total abuse potential score, with higher scores indicating higher abuse potential.

SECONDARY OUTCOMES:
Change from Baseline in score on Child Behavior Checklist (CBCL) at 6 months | Baseline and 6 months
  The CBCL uses a 3-point response scale (not true to very true) to assess child internalizing and externalizing symptoms (mental health symptoms)
Change from Baseline in score on Child Behavior Checklist (CBCL) at 18 months | Baseline and 18 months
  The CBCL uses a 3-point response scale (not true to very true) to assess child internalizing and externalizing symptoms (mental health symptoms)
Change from Baseline in scores on Parenting Stress Index at 6 months | Baseline and 6 months
  The PSI includes 36 items assessing parent-child dysfunctional interaction, parental distress and perceptions of a difficult child.
Change from Baseline in scores on Parenting Stress Index at 18 months | Baseline and 18 months
  The PSI includes 36 items assessing parent-child dysfunctional interaction, parental distress and perceptions of a difficult child.
Change from Baseline in score on Childhood injuries at 6 months | Baseline and 6 months
  Mothers will report on the type and severity of children's injuries that occurred in the home during the past 6-months.
Change from Baseline in score on Childhood injuries at 18 months | Baseline and 18 months
  Mothers will report on the type and severity of children's injuries that occurred in the home during the past 6-months.
Change from Baseline in score on Child Quality of Life at 6 months | Baseline and 6 months
  The parent-report version of of the Child Health Utility measure (CHU9D) will assess children's health-related quality of life.
Change from Baseline in score on Child Quality of Life at 18 months | Baseline and 18 months
  The parent-report version of of the Child Health Utility measure (CHU9D) will assess children's health-related quality of life.
Change from Baseline in score on Parent Quality of Life at 6 months | Baseline and 6 months
  The parent will self-report their quality of life using the EQ-5D-5L utility index.
Change from Baseline in score on Parent Quality of Life at 18 months | Baseline and 18 months
  The parent will self-report their quality of life using the EQ-5D-5L utility index.

OTHER OUTCOMES:
Client satisfaction | Up to 12 weeks
  Satisfaction survey of parents' view of SafeCare Kenya services
Provider fidelity | Up to 30 months
  Assessment of Provider's delivery of SafeCare Kenya sessions
Parent Interview | Up to 4 months
  Interview protocol to learn what parents liked and did not like about SafeCare Kenya, changes they suggest, and benefit to future families
Provider Interview | Up to 30 months
  Interview protocol to learn what providers liked and did not like about SafeCare Kenya, changes they suggest, benefit to future families, value and challenges with delivery modalities, value and challenges with training and coaching support
Trainer Interview | Up to 30 months
  Interview protocol to learn what trainers liked and did not like about SafeCare Kenya, changes they suggest, benefit to future families, value and challenges with delivery modalities, value and challenges with training and coaching
Stakeholder Interview | Up to 30 months
  Interview protocol to learn what stakeholders liked and did not like about SafeCare Kenya and its implementation, along with suggested changes
Readiness Assessment for the Prevention of Child Maltreatment (RAP-CM) | Up to 30 months
  WHO Survey about a country's preparedness to implement a child maltreatment prevention program

CONTACTS AND LOCATIONS:
Overall Officials: Jenelle R. Shanley, PhD, Principal Investigator — Pacific University; David Ndetei, MD, Principal Investigator — Africa Institute of Mental and Brain Health; Lisa P. Armistead, PhD, Principal Investigator — Georgia State University
Locations (1):
- Africa Institute of Mental and Brain Health, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No